CLINICAL TRIAL: NCT02767440
Title: Families on Track: A Digital Health Behavioral Intervention for Parents Seeking Treatment for Their Child With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00072648
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Childhood Obesity; Hypertension; Diabetes; Dyslipidemia
MeSH Terms: conditions — Obesity; Pediatric Obesity; Hypertension; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Families on Track Intervention (Experimental): This is a pre-post study. Enrolled parents will receive the Families on Track intervention plus usual care at the Healthy Lifestyles clinic at Duke University.
  Interventions: Behavioral: Families on Track Intervention

INTERVENTIONS:
Behavioral: Families on Track Intervention — Parents will receive the standard of care activities at the Healthy Lifestyles clinic at Duke University. They will also receive a modified version of the previously conducted Track intervention, a digital health weight loss intervention for adults in community health centers . The intervention will utilize the Interactive Obesity Treatment Approach (iOTA). iOTA uses a computer algorithm to assign 3 personalized behavioral goals known to create an energy deficit to produce weight loss (e.g., sugary drinks, fast food consumption walk 10,000 steps/day, etc). Participants will track these goals via interactive voice response (IVR) and text messaging technologies each week. They will receive immediate feedback based on self-monitoring data and skills training videos to learn how to make the behavioral changes necessary for weight loss. Intervention participants will also receive an analog bathroom scale and a pedometer to self-monitor daily weights and steps.

SUMMARY:
Current models of outpatient childhood obesity treatment focus on the child's health habits, with limited efficacy. In part, this may be because childhood obesity is highly sensitive to parental lifestyle habits, who are often not a direct target of child obesity interventions. This study aims to target weight loss among overweight parents of 2-16 year old children with obesity enrolled in the Duke Healthy Lifestyles Program (HL) in order to augment child body mass index reduction. The intervention, " Families on Track" is a digital health intervention platform using the Interactive Obesity Treatment Approach (iOTA).

DETAILED DESCRIPTION:
Parents in the program will receive the family-based treatment protocol provided by the Healthy Lifestyles clinic. First, families attend a half-day session at the clinic where child anthropometrics and labs are obtained, and nutrition and physical activity group counseling is provided. Height and weight of the primary adult caregiver are measured and BMI is calculated. Second, families return 2 weeks later to meet individually with a pediatric obesity medical provider and a registered dietitian. Thereafter, frequency of visits is determined based on the families needs with a final visit 1 year after starting treatment. The ideal is to have visits with the HL staff at intervals of 4-6 weeks for 5 more visits to complete the primary phase of the program over 6 months.

Parents enrolled in the study will also receive the Track intervention. The investigators will use a modified version of the Track intervention, which utilized the Interactive Obesity Treatment Approach (iOTA). iOTA uses a computer algorithm to assign 3-4 personalized behavioral goals known to create an energy deficit to produce weight loss (e.g., sugary drinks, fast food consumption walk 10,000 steps/day, etc). The team at Duke Digital Health has shown that iOTA can be successfully delivered to adults on multiple modalities -- web, text messaging and interactive voice response phone calls. Each week, participants will receive a prompt from the Track intervention system in order to self-monitoring these behaviors goals. These prompts will be delivered either via interactive voice response or text message. Intervention participants will also receive an analog bathroom scale and a pedometer to self-monitor daily weights and steps.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years
* BMI: 25-50 kg/m2
* English speaking
* Mobile phone ownership
* Willingness to send and receive multiple text messages/day
* living in the same household as a Healthy Lifestyles patient ages 2-16

Exclusion Criteria:

* Current pregnancy or lactation
* Prior or planned bariatric surgery Both child and parent participation in other obesity trials - including the evaluation of the Bull City Fit Program at the Healthy Lifestyles program
* History of heart attack, stroke, bipolar disorder schizophrenia or recent cancer diagnosis
* Plans to relocate within 1 year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
change in parent weight over 6 months | baseline, 6 months

SECONDARY OUTCOMES:
change in parent BMI over 6 months | baseline, 6 months
change in parent waist circumference over 6 months | baseline, 6 months
change in parent blood pressure over 6 months | baseline, 6 months
change in child lipid panel (total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides) over 6 months | baseline, 6 months
change in child glucose, insulin, and HbA1c over 6 months | baseline, 6 months
change in child z-BMI over 6 months | baseline, 6 months
change in child blood pressure over 6 months | baseline, 6 months
change in child cardiovascular fitness/physical conditioning | baseline, 6 months
  measured by 3-minute step test, 1-minute recovery heart rate over 6 months
change in parent diet over 6 months | baseline, 6 months
  as measured by a Food Frequency Questionnaire
change in parent exercise behaviors over 6 months | baseline, 6 months
  as measured by Paffenbarger Exercise Habits Questionnaire
change in child consumption of sugar sweetened beverages over 6 months | baseline, 6 months
  as measured by a Food Frequency Questionnaire
change in child consumption of fruits and vegetables over 6 months | baseline, 6 months
  as measured by a Food Frequency Questionnaire
change in child consumption of sugary snacks over 6 months | baseline, 6 months
  as measured by a Food Frequency Questionnaire
change in child number of minutes of physical activity | baseline, 6 months
  measured by the Physical Activity Questionnaire for Children
change in child number of minutes of screen time | baseline, 6 months
  measured by the Physical Activity Questionnaire for Children
change in parent depression over 6 months | baseline, 6 months
  measured by Patient Health Questionnaire (PHQ-8)
change in child quality of life over 6 months | baseline, 6 months
  measured by Sizing Me Up sub-scales
change in child perceived healthy eating and physical activity social/environmental support over 6 months | baseline, 6 months
change in parent perceived healthy eating and physical activity social/environmental support over 6 months | baseline, 6 months
change in home food environment over 6 months | baseline, 6 months
  measured by Home Food Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Armstrong, MD, Principal Investigator — Duke University Health System, Duke Healthy Lifestyles; Dori M Steinberg, PhD, RD, Principal Investigator — Duke University
Locations (1):
- Duke Pediatrics Healthy Lifestyles Clinic, Durham, NC, North Carolina, United States